CLINICAL TRIAL: NCT07135427
Title: Genetic Variation in IgG as a Mechanism for Immune Deficiency and Exacerbations in AATD
Brief Title: Genetic Variation in IgG in Alpha 1 Antitrypsin Deficiency
Acronym: IgG in AATD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Alpha-1 Foundation (Other)
Responsible Party: Principal Investigator, David Lafon, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB300008528(000547878); Research award (Other: Alpha-1 Foundation)
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-08

CONDITIONS: Alpha 1-Antitrypsin; COPD; Antibody Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SERPINA1 'Z' heterozygotes (Experimental): Participants who are heterozygous for the SERPINA1 'Z' allele with either 0 or 2+ exacerbations in the previous year, and have not received pneumococcal vaccination within 5 years will be given PCV20.
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 20-valent pneumococcal conjugate vaccine — Administration of PCV20

SUMMARY:
The goal of this study is to learn whether patients who have a genetic mutation in the genes that cause alpha 1 antitrypsin deficiency also have genetic variation in nearby genes that can increase risk for reduced immune function and respiratory infections.

To investigate this hypothesis, we will compare immune responses to the 20-valent pneumococcal conjugate vaccine (PCV20, Pfizer) between participants who have one abnormal copy of the SERPINA1 gene and either no COPD exacerbations, vs those with 2 or more COPD exacerbations in the past year.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are heterozygous for a SERPINA1 Z allele
* Have either had no COPD exacerbations or 2 or more exacerbations in the previous year
* Has not received a pneumococcal conjugate vaccine within the past 5 years, or has only received the pneumococcal polysaccharide vaccine in the past

Exclusion Criteria:

* Received a pneumococcal conjugate vaccine within the past 5 years
* Known allergy, severe adverse reaction, or other sensitivity to pneumococcal conjugate vaccines

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Antibody response | 4 weeks from baseline measurement
  Pneumococcal antibody levels/function, total IgG levels, IgG subclass levels; magnitude of change from baseline

SECONDARY OUTCOMES:
Lymphocyte profile | Baseline, 4 weeks post-vaccination
  B and T cell lymphocyte subsets

OTHER OUTCOMES:
Gene variants | Baseline
  Variants in SERPINA1, IGHG genes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided